CLINICAL TRIAL: NCT04311944
Title: Early Fast-Track Versus Standard Care for Persons With HIV Initiating Tenofovir Disoproxil Fumarate-Lamivudine-Dolutegravir (TLD) in Haiti: A Pilot Randomized Trial
Brief Title: Early Fast-Track Versus Standard Care for Persons With HIV Initiating TLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other)
Collaborators: Brigham and Women's Hospital (Other); Weill Medical College of Cornell University (Other); Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 212336
Record Dates: First submitted 2020-03-15; First posted 2020-03-17 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: HIV-1-infection
Keywords: HIV; Antiretroviral therapy; Differentiated care; Expedited services

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to early fast-track vs. standard care.
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early Fast-Track Care (Experimental): Participants will be eligible for fast-track care after 8 to 12 weeks, if viral load is suppressed (<200 copies/mL)
  Interventions: Other: Early fast-track care
- Standard (Deferred Fast-track) Care (Active Comparator): Participants will be eligible for fast-track care after 24 weeks, if viral load is suppressed (<200 weeks)
  Interventions: Other: Standard (deferred fast-track) care

INTERVENTIONS:
Other: Early fast-track care — Participants will be eligible for fast-track care at 8 weeks if their HIV-1 RNA is <200 copies/mL and they meet other eligibility criteria. If HIV-1 RNA is 200 copies/mL or higher at 8 weeks, then it will be repeated at 12 weeks, and those with HIV-1 RNA <200 copies will then be eligible for fast-track care, if they meet other eligibility criteria.
  Arms: Early Fast-Track Care
Other: Standard (deferred fast-track) care — Participants will be eligible for fast-track care at 24 weeks, if their HIV-1 RNA is <200 copies.mL, and they meet other eligibility criteria.
  Arms: Standard (Deferred Fast-track) Care

SUMMARY:
This study will evaluate the clinical efficacy of using earlier fast-track services compared to the standard of care in a clinical setting to improve retention in care and virologic suppression for patients who are initiating a dolutegravir-based antiretroviral therapy regimen.

DETAILED DESCRIPTION:
With current approaches to HIV care, patients generally do not qualify for expedited services until they have been in care for 6 to 12 months. Once they have achieved an undetectable viral load and/or high adherence, patients qualify for expedited services with fewer clinic visits. The problem with this approach is that it's time-intensive early in ART care, when attrition rates are highest. A potential solution to this problem is to provide earlier fast-track care for patients on dolutegravir-based regimens with viral suppression. This strategy is feasible due to the high potency and rapid declines in viral load with dolutegravir-based regimens.

We will compare a strategy of early fast-track care (8 to 12 weeks, for patients with viral suppression) versus standard initiation of fast-track care (after 6 months in care, with viral suppression). All participants will receive the same ART regimen, the combination regimen of Tenofovir Disoproxil Fumarate-Lamivudine-Dolutegravir.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of positive HIV status (test conducted at GHESKIO)
* Age ≥18 years of age
* Eligible for TLD regimen, according to Haitian Ministry of Health guidelines
* Initiate ART within 3 days prior to enrollment
* Lives in Port-au-Prince metropolitan area
* Ability and willingness to give written informed consent
* Use of reliable contraception (for women of childbearing potential);
* Physician-confirmed WHO Stage 1 or 2 disease

Exclusion Criteria:

* Not ART-naïve (history of ART for any duration in the past)
* World Health Organization Stage 3 or 4 disease;
* Pregnancy or breastfeeding at the screening visit;
* Planning to become pregnant during the study period;
* Active drug, alcohol use, or mental condition that would interfere with the ability to adhere to study requirements, in the opinion of the study physician;
* Creatinine clearance (CrCl) <50 within 1 month prior to study entry;
* ALT and/or AST> 5X upper limit of normal (ULN) within 1 month prior to study entry;
* Planning to transfer care to another clinic during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-29 (Estimated)

PRIMARY OUTCOMES:
Viral suppression - 200 copies/mL cut-off | 48 weeks after study enrollment
  Proportion of participants with HIV-1 RNA <200 copies/mL

SECONDARY OUTCOMES:
Viral suppression - 50 copies/mL cut-off | 48 weeks after study enrollment
  Proportion of participants with HIV-1 RNA <50 copies/mL
Viral suppression - 1000 copies/mL cut-off | 48 weeks after study enrollment
  Proportion of participants with HIV-1 RNA <1000 copies/mL
Adherence of at least 90% | 48 weeks after enrollment
  Adherence to antiretroviral therapy of at least 90% as measured by pharmacy refill records
Medication tolerability | 48 weeks after enrollment
  Proportion of participants discontinuing tenofovir disoproxil/lamivudine/dolutegravir regimen
Cost | 48 weeks after enrollment
  Total cost of early fast-track and standard (deferred fast-track) care from the health center perspective
Time in clinic | 48 weeks after enrollment
  Median time in clinic

CONTACTS AND LOCATIONS:
Overall Officials: Colette Guiteau, MD, Principal Investigator — Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic; Serena Koenig, MD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the end of the study.
Supporting Information: Study Protocol, CSR
Time Frame: Within 48 weeks after study completion
Access Criteria: Open access